CLINICAL TRIAL: NCT02004704
Title: A Long-Term Study to Assess the Ongoing Safety and Efficacy of Olipudase Alfa in Patients With Acid Sphingomyelinase Deficiency
Brief Title: A Long-Term Study of Olipudase Alfa in Patients With Acid Sphingomyelinase Deficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS13632; 2013-000051-40 (EudraCT Number)
Expanded Access: NCT04877132 (Approved for marketing)
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Sphingomyelin Lipidosis
MeSH Terms: conditions — Niemann-Pick Disease, Type A | interventions — olipudase alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GZ402665 (Experimental): GZ402665 administered intravenously once every 2 weeks at the dose each participant was receiving at the end of their previous olipudase alfa study, for 9 years or until olipudase alfa becomes commercially accessible, whichever comes first, unless the participant decides to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa is commercially accessible.
  Interventions: Drug: GZ402665

INTERVENTIONS:
Drug: GZ402665 — Pharmaceutical form: Powder for concentrate for solution for infusion
  Route of administration: intravenous infusion
  Other Names: Olipudase alfa

SUMMARY:
The primary objective of this study was to obtain data regarding the safety of olipudase alfa in participants with acid sphingomyelinase deficiency (ASMD) who were exposed to long term treatment with olipudase alfa.

The secondary objectives of this study were to obtain data regarding the efficacy of olipudase alfa and to characterize olipudase alfa pharmacodynamics (PD) and pharmacokinetics (PK) following long-term administration.

DETAILED DESCRIPTION:
LTS13632 is a multicenter, nonrandomized, open-label, long-term extension study of participants with ASMD who have previously participated in a study of olipudase alfa. (DFI13803 for pediatric participants and DFI13412 for adult participants).

The maximum study duration per participant was 9 years or until olipudase alfa becomes commercially accessible. Notwithstanding the above, every pediatric participant were treated in LTS13632 study for at least 3 years to comply with the requirements agreed in the olipudase alfa Pediatric Investigational Plan.

ELIGIBILITY:
Inclusion criteria:

* The participant completed the treatment period of a previous study of olipudase alfa with an acceptable safety profile in the opinion of the investigator and sponsor.
* The participant and/or the participant's parent(s)/legal guardian(s) was willing and able to provide signed written informed consent.
* The participant who is female and of childbearing potential must have had a negative urine pregnancy test for beta human chorionic gonadotropin (β HCG).
* Female participants of childbearing potential and sexually mature male participants must have been willing to practice true abstinence in line with their preferred and usual lifestyle or use 2 acceptable effective methods of contraception up to 15 days following their last dose of study drug.

Exclusion criteria:

* The participant had any new condition or worsening of an existing condition which in the opinion of the investigator would make the participant unsuitable for enrollment, or could interfere with the participation or completion the study.
* The participant, in the opinion of the investigator, was unable to adhere to the requirements of the study.
* The participant was unwilling or unable to abstain from the use of alcohol for 1 day prior to and 3 days after each olipudase alfa infusion for the duration of the treatment period.
* The participant was unwilling or unable to avoid, for 10 days before and 3 days after liver biopsies, medications or herbal supplements that are potentially hepatotoxic (only participants who previously participated in the DFI13412 study).
* The participant required medication(s) that may decrease olipudase alfa activity (eg, fluoxetine, chlorpromazine; tricyclic antidepressants [eg, imipramine, desipramine]).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (9):
- Investigational Site Number 840001, New York, New York, United States
- Investigational Site Number 056001, Leuven, Belgium
- Investigational Site Number 076001, Porto Alegre, Brazil
- Investigational Site Number 250002, Bron, France
- Investigational Site Number 276002, Hochheim am Main, Germany
- Italy (2):
  - Investigational Site Number 380002, Sassari
  - Investigational Site Number 380001, Udine
- United Kingdom (2):
  - Investigational Site Number 826001, London
  - Investigational Site Number 826002, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Scarpa M, Diaz GA, Giugliani R, Jones SA, Mengel E, Guffon N, Witters P, Ganesh J, Armstrong NM, Srivastava S, Kim Y. Long-Term Safety and Clinical Outcomes With Olipudase Alfa Enzyme Replacement Therapy in Children and Adolescents With Acid Sphingomyelinase Deficiency. J Inherit Metab Dis. 2025 Sep;48(5):e70086. doi: 10.1002/jimd.70086. PMID 40937531
- [Derived] Thurberg BL, Diaz GA, Lachmann RH, Schiano T, Wasserstein MP, Ji AJ, Zaher A, Peterschmitt MJ. Long-term efficacy of olipudase alfa in adults with acid sphingomyelinase deficiency (ASMD): Further clearance of hepatic sphingomyelin is associated with additional improvements in pro- and anti-atherogenic lipid profiles after 42 months of treatment. Mol Genet Metab. 2020 Sep-Oct;131(1-2):245-252. doi: 10.1016/j.ymgme.2020.06.010. Epub 2020 Jun 24. PMID 32620536
- [Derived] Wasserstein MP, Diaz GA, Lachmann RH, Jouvin MH, Nandy I, Ji AJ, Puga AC. Olipudase alfa for treatment of acid sphingomyelinase deficiency (ASMD): safety and efficacy in adults treated for 30 months. J Inherit Metab Dis. 2018 Sep;41(5):829-838. doi: 10.1007/s10545-017-0123-6. Epub 2018 Jan 5. PMID 29305734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 9 investigational sites in 6 countries between 04 Dec 2013 and 06 Sep 2023.
Pre-assignment Details: A total of 25 participants (5 adult participants from study DFI13412 [NCT01722526] and 20 pediatric participants from study DFI13803 [NCT02292654]) directly rolled over and continued treatment in this study.
Groups:
- Olipudase Alfa: Participants From DFI13412 (Adults): Participants continued to receive olipudase alfa at the same dose as at the completion of original study- DFI13412 (up to 3.0 milligram/kilogram [mg/kg]) via intravenous (IV) infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible.
- Olipudase Alfa: Participants From DFI13803 (Pediatrics): Participants continued to receive olipudase alfa at the same dose as at the completion of original study- DFI13803 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible. During the study, pediatric participants who reached adult age (18 years old) received the adult infusion volume.
Period: Overall Study
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Started | 5 | 20
Completed | 5 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set consisted of all enrolled participants who received at least 1 infusion (partial or total) of olipudase alfa in the current study.
Groups:
- Olipudase Alfa: Participants From DFI13412 (Adults): Participants continued to receive olipudase alfa at the same dose as at the completion of original study- DFI13412 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible.
- Total: Total of all reporting groups
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics) | Total
Number analyzed (Participants) | 5 | 20 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.25) | 7.6 (4.43) | 12.5 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 3 | 10 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 17 | 22
  Other | 0 | 1 | 1
  Southeast Asian | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs) and Adverse Events of Special Interest (AESIs) Except Infusion-Associated Reactions (IARs)
Description: An AE: Any untoward medical occurrence in participant or clinical investigation participant administered with pharmaceutical product, which did not necessarily have to have causal relationship with study treatment. SAEs: Any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization/prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was congenital anomaly/birth defect, was medically important event. TEAEs: AEs that started during on-treatment period-either in this study or in original study which were ongoing at the time the participant signed the written informed consent. An AESI: AE (serious or nonserious) of scientific and medical concern specific to sponsor's product or program, for which ongoing monitoring and rapid communication by investigator to sponsor was appropriate.
Time Frame: From the signature of informed consent up to 9 years or until olipudase alfa was commercially accessible, whichever came first
Population: Results are based on the Safety analysis set which consisted of all enrolled participants who received at least 1 infusion (partial or total) of olipudase alfa in the current study.
Measure: Count of Participants; unit: Participants
Groups:
- Olipudase Alfa: Participants From DFI13803 (Pediatrics): Participants continued to receive olipudase alfa at the same dose as the completion of original study- DFI13803 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible. During the study, pediatric participants who reached adult age (18 years old) received the adult infusion volume.
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  Any TEAE | 5 | 20
  Any TESAE | 1 | 10
  AESI: Any Pregnancies | 0 | 0
  AESI: Symptomatic Overdose | 0 | 0
  AESI: Dose-limiting toxicities | 0 | 10
  Any TEAEs leading to treatment discontinuation | 0 | 0
  Any TEAEs leading to death | 0 | 0

2. Primary Outcome: Number of Participants With IARs
Description: Protocol-defined IARs were AEs that occurred during the infusion or within up to 24 hours after the start of infusion and were considered as related or possibly related to the study treatment by the investigator or the sponsor. Events occurring greater than or equal to (>=) 24 hours after the start of an infusion might have been judged an IAR at the discretion of the investigator or sponsor. Algorithm-defined IARs were all AEs that started between the start of infusion and the end of infusion plus 24 hours, irrespective of the perceived relation with study treatment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  Protocol-defined IARs | 4 | 13
  Algorithm-defined IARs | 5 | 20

3. Primary Outcome: For Adults: Number of Participants With Abnormality in Complete Physical Examinations Including Abbreviated Physical Exam
Description: A complete physical examination included assessment of the participant's general appearance, general neurological status, skin, head, eyes, ears, nose, throat, lymph nodes, heart, lungs, abdomen, and extremities/joints. Shift from Baseline was monitored. An abbreviated physical exam (general appearance only) was only performed pre- and post-infusion for those who did not do complete exam.
Time Frame: Baseline (Day 1 of original study), Month 78
Population: Results are based on the Safety analysis set which consisted of all enrolled participants who received at least 1 infusion (partial or total) of olipudase alfa in the current study. Only those participants with data collected at specified timepoints are reported.
Measure: Count of Participants; unit: Participants
Groups:
- Olipudase Alfa: Participants From DFI13412 (Adults): Participants continued to receive olipudase alfa as at the same dose as at the completion of original study- DFI13412 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible.
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults)
Number analyzed (Participants) | 5
Participants
  General Appearance | 0
  General Neurological Status | 0
  Skin | 1
  Head, Eyes, Ears, Nose and Throat | 1
  Lymph Nodes | 0
  Heart | 0
  Lungs | 0
  Abdomen | 1
  Extremities/Joints | 0
  Abbreviated Physical Exam | 0

4. Primary Outcome: For Pediatrics: Number of Participants With Abnormality in Complete Physical Examinations Including Abbreviated Physical Exam
Description: A complete physical examination included assessment of the participant's general appearance, skin, head, eyes, ears, nose, throat, lymph nodes, heart, lungs, abdomen, and extremities/joints. Shift from Baseline was monitored. An abbreviated physical exam (general appearance only) was only performed pre- and post-infusion for those who did not do complete exam.
Time Frame: Baseline (Day 1 of original study), Month 84
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5
Participants
  General Appearance | 0
  Skin | 1
  Head, Eyes, Ears, Nose and Throat | 0
  Lymph Nodes | 0
  Heart | 0
  Lungs | 0
  Abdomen | 2
  Extremities/Joints | 0
  Abbreviated Physical Exam | 0

5. Primary Outcome: For Adults: Number of Participants With Abnormality in Extended Neurological Examinations
Description: Extended neurological examination for adults included examination of mental status. Shift from Baseline was monitored.
Time Frame: Baseline (Day 1 of original study), Month 78
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults)
Number analyzed (Participants) | 5
Participants | 0

6. Primary Outcome: For Pediatrics: Number of Participants With Abnormality in Extended Neurological Examinations
Description: The neurological examination in pediatric participants included examination of mental status, cranial nerve examination, motor examination: tone, reflexes examination, sensory examination, coordination, gait and coordination, and strength examination. Shift from Baseline was monitored.
Time Frame: Baseline (Day 1 of original study), Month 84
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5
Participants
  Mental Status | 0
  Cranial Nerve Examination | 0
  Motor Examination: Tone | 0
  Reflexes Examination | 0
  Sensory Examination | 0
  Coordination | 0
  Gait and Coordination | 0
  Strength Examination | 0

7. Primary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities (PCSA) in Vital Signs
Description: PCSA: Heart Rate: High: >=120 beats per minute (bpm) (adults [ad], adolescents [ado], children [chi]), >=140 bpm (early chi [ec]), >=175 bpm (infants[inf]) & increase from baseline (IFB)>=20 bpm for all age ranges (AAR), HR Low: <=50 bpm (ad, ado, chi), <=75 bpm (ec), <=80 bpm (inf) & decrease from baseline (DFB) >=20 bpm for AAR. Systolic blood pressure: High: >= 160 millimeters of mercury (mmHg) (ad); >=119 mmHg (ado), >=108 mmHg (chi), >=101 mmHg (ec),>=98 mmHg (inf) & IFB >=20 mmHg for AAR. SBP Low: <=95 mmHg (ad), <=90 mmHg (ado), <= 80mm Hg (chi), <=70 mmHg (ec), <=70 mmHg (inf) & DFB >=20 mmHg for AAR. Diastolic blood pressure: High:>110 mmHg (ad), >=78 mmHg (ado), >=72 mmHg (chi), >=59 mmHg (ec), >=54 mmHg (inf) and IFB >=10 mmHg for AAR. DBP Low:<=45 mmHg (ad), <=54 mmHg (ado), <=48 mmHg (chi), <=34mmHg (ec and inf) & DFB>=10 mmHg for AAR.
Time Frame: Baseline (Day 1 of original study) up to 9 years or until olipudase alfa was commercially accessible, whichever came first
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  Heart Rate: High | 1 | 9
  Heart Rate: Low | 2 | 10
  Systolic blood pressure: High | 2 | 16
  Systolic blood pressure: Low | 5 | 11
  Diastolic blood pressure: High | 0 | 19
  Diastolic blood pressure: Low | 5 | 19

8. Primary Outcome: Number of Participants With PCSA in Clinical Chemistry Parameters
Description: PCSA: Creatinine High, category 1: >=150 micromole/L (umol) (adults), >=132 umol/L or 1.5 mg/deciliter (dL) (adolescents), >=90 umol/litre (L) or 1.1 mg/dL (children), >53 umol/L or 0.6 mg/dL (early children and infants); category 2: >=30% IFB (adults). Blood Urea Nitrogen: >=17 millimole (mmol)/L (adults), >=6.4 mmol/L or 18 mg/dL (pediatrics [ped]). Glucose Low<=3.9 mmol/L and <lower limit of normal (adults), <2.7 mmol/L (ped), High: >=11.1 mmol/L (unfasted), >7 mmol/L (fasted) (adults), >=7 mmol/L (fasted after >12 hours of fast); >=10.0 mmol/L (unfasted) (ped).
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  Creatinine: High, category 1 | 0 | 0
  Creatinine: High, category 2 | 1 | 4
  Blood Urea Nitrogen: High | 0 | 15
  Glucose: Low | 5 | 2
  Glucose: High | 1 | 0

9. Primary Outcome: Number of Participants With PCSA in Liver Function Tests
Description: PCSA: Alanine aminotransferase (ALT) >3 x upper limit of normal (ULN). Aspartate aminotransferase (AST) >3 x ULN. Alkaline phosphatase (ALP) > 1.5 x ULN. Total Bilirubin >1.5 x ULN (ad) and >1.3 x ULN (ped). ALT and total bilirubin: ALT > 3 x ULN and total bilirubin > 2 x ULN.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  ALT | 0 | 5
  AST | 0 | 6
  ALP | 0 | 5
  Total Bilirubin | 3 | 1
  ALT and Total Bilirubin | 0 | 0

10. Primary Outcome: Number of Participants With PCSA in Hematology Parameters
Description: PCSA: White blood cells (WBC): Low: <3.0 Giga (G)/L (Non-Black [NB])/<2.0 G/L (Black [B])(ad), <4.5 G/L (ado), <5.0 G/L(chi), <3.0 G/L (ec), <4.0 G/L (inf), High: >=16.0 G/L(ad), >13.5 G/L (ado), >17.0 G/L(chi), >16 G/L (ec), >20 G/L (inf). Hemoglobin-ad: Low-1: <=115 g/dL (Male [M])/<=95 g/dL (Female [F]), 20% DFB for both, High:>=185 g/L (M)/>=165 g/L (F), Low-2: DFB>=20 g/L (ad), <10 g/dL (ado, chi, ec); <9.0 g/dL (inf); 20% DFB for all. Platelets: Low: <100 G/L (AAR) and 20% DFB and High: >=700 G/L (ad and ped).
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  WBC: Low | 2 | 16
  WBC: High | 0 | 0
  Hemoglobin: Low-1 | 0 | 0
  Hemoglobin: High | 1 | 0
  Hemoglobin: Low-2 | 2 | 0
  Platelets: Low | 2 | 7
  Platelets: High | 0 | 0

11. Primary Outcome: Number of Participants With PCSA in Electrocardiogram (ECG)
Description: PCSA: Heart rate: High:>=120 bpm (ad, ado, chi), >=140 bpm (ec), >=175 bpm (inf) & IFB>=20 bpm for AAR, Heart rate: Low: <=50 bpm (ad, ado, chi), <=75 bpm (ec), <=80 bpm (inf) & DFB >=20 bpm for AAR. PR duration: High: >=200 milliseconds (ms) (ad) and IFB>=20 ms, >180 ms (ado), 170 ms (chi), 160 ms (ec), and 140 ms (inf). QT correction-Bazett (QTcB): Borderline absolute (category 1): 431-450 ms (ad and ado M, chi, ec and inf), 451-470 ms (ad and ado F), Prolonged-absolute (category 2): >450 ms (ad and ado M and chi, ec and inf), >470 ms (ad and ado F), Additional-absolute (category 3): >=500 ms (AAR), Borderline increase (category 4): 30-60 ms (AAR), Prolonged increase (category 5): > 60 ms (AAR).
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  Heart rate: High | 0 | 3
  Heart rate: Low | 1 | 2
  PR duration: High | 0 | 6
  QTcB: Category 1 | 5 | 13
  QTcB: Category 2 | 5 | 8
  QTcB: Category 3 | 0 | 0
  QTcB: Category 4 | 5 | 7
  QTcB: Category 5 | 2 | 1

12. Primary Outcome: For Adults: Percent Change From Baseline in Pre-Infusion Plasma Ceramide at Month 90
Description: Plasma samples were collected to evaluate ceramide levels for safety biomarker analysis. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 90 (pre-infusion)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults)
Number analyzed (Participants) | 4
percent change | -65.66 (12.58)

13. Primary Outcome: For Pediatrics: Percent Change From Baseline in Pre-Infusion Plasma Ceramide at Month 66
Description: as for outcome 12
Time Frame: Baseline (Day 1 of original study) and Month 66 (pre-infusion)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5
percent change | -69.16 (10.04)

14. Primary Outcome: Participants From Adult Study DFI13412: Number of Participants With Abnormal Liver Biopsy
Description: Liver biopsy samples were evaluated for sphingomyelin accumulation and liver pathology in the participants who previously participated in the DFI13412 study who were at least 18 years old when they entered in this study. Sphingomyelin accumulation was quantified in liver by computer morphometry of high-resolution light microscopy images. Fibrosis grading was assessed on the Laennec scoring system, which grades the extent of fibrosis on a scale from 0 to 4 (0=none; 1=minimal; 2=mild; 3=moderate; 4=cirrhosis). Higher score indicated more severity.
Time Frame: Baseline (Day 1 of original study) and Month 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults)
Number analyzed (Participants) | 5
Participants
  Baseline: Stage 0 | 1
  Baseline: Stage 1 | 1
  Baseline: Stage 2 | 2
  Baseline: Stage 3 | 1
  Baseline: Stage 4 | 0
  Month 36: Stage 0 | 0
  Month 36: Stage 1 | 1
  Month 36: Stage 2 | 1
  Month 36: Stage 3 | 2
  Month 36: Stage 4 | 1

15. Primary Outcome: Participants From Pediatric Study DFI13803: Number of Participants With Abnormalities in Liver Ultrasound Doppler
Description: Liver ultrasound doppler was performed for pediatric participants transitioning from DFI13803 to document hepatic blood flow characteristics, principally portal vein pressure, and blood flow direction. The parameters evaluated were liver dysmorphic findings, liver surface abnormalities, mild ascites and hepatic steatosis. Liver ultrasound Doppler was performed using methods that were compatible with the standard institutional procedures of the investigational site.
Time Frame: Baseline (Day 1 of original study), Week 2 and Months 12, 18 and 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 20
Participants
  Liver dysmorphic findings: Baseline | 6
  Liver dysmorphic findings: Month 12 | 3
  Liver dysmorphic findings: Month 18 | 1
  Liver dysmorphic findings: Month 24 | 0
  Liver surface abnormalities: Baseline | 5
  Liver surface abnormalities: Month 12 | 0
  Mild ascites: Baseline | 3
  Mild ascites: Week 2 | 2
  Mild ascites: Month 12 | 0
  Hepatic steatosis: Baseline | 1
  Hepatic steatosis: Month 12 | 0

16. Primary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) Against Olipudase Alfa
Description: Blood samples were collected for the presence of ADAs against olipudase alfa. Treatment-boosted ADA: Positive ADA status positive at baseline (pre-existing ADA) and ADA titer level anytime post-baseline significantly higher than that at baseline. Transient ADA: Treatment-induced ADA detected only at 1 sampling time point post-baseline and treatment-induced ADA detected at 2 or more sampling time points post-baseline, where first and last ADA-positive samples (irrespective of any negative samples in between) separated by period of less than 16 weeks, and participant's last sampling time point was ADA-negative. Persistent ADA response: Treatment-induced ADA detected at 2 or more sampling time points post-baseline, where first and the last ADA-positive on-treatment sample (irrespective of any negative samples in between) separated by at least 16 weeks. Treatment-induced: ADA detected in the last 2 sampling time points, irrespective of the time period in between.
Time Frame: as for outcome 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 20
Participants
  ADA positive at baseline | 0 | 2
  Treatment-boosted ADAs | 0 | 1
  Treatment-induced ADAs | 3 | 14
  Transient ADA response | 0 | 1
  Indeterminate ADA response | 0 | 0
  Persistent ADA response | 3 | 12
  ADA positive since first dose of olipudase alfa | 3 | 15
  Treatment-emergent ADA | 3 | 15

17. Secondary Outcome: Percent Change From Baseline in Spleen and Liver Volumes at Month 102 for Adults and Month 84 for Pediatrics
Description: Spleen and liver volumes were assessed by abdominal magnetic resonance imaging (MRI) collected and read centrally by a third party blinded to participant number and study visit to quantify the degree of splenomegaly and hepatomegaly at specified time points. Spleen/Liver volume in multiples of normal (MN) = Spleen/Liver volume (cubic centimeter [cm^3]) / [2xweight (kg)] where weight was the available value closest to the MRI scan date. Negative value signifies reduction of volume. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study), Month 102 for adults and Month 84 for pediatrics
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 7
percent change
  Spleen volume | -63.60 (6.34) | -75.56 (7.15)
  Liver volume | -46.71 (14.40) | -59.55 (14.26)

18. Secondary Outcome: Change From Baseline in Pulmonary Imaging by High Resolution Computed Tomography (HRCT) at Month 102 for Adults and Month 84 for Pediatrics
Description: Pulmonary imaging of chest using HRCT was obtained for qualitative assessment of ground glass appearance, interstitial lung disease, pleural thickening and reticulo-nodular density. Images were collected and read centrally by a third party blinded to participant number and study visit. Lung fields were scored subjectively for degree of diffuse lung disease (infiltrative lung disease) in scale of 0-3 ranging from 0 = No disease, 1 = Mild (affecting 1% to 25% of the lung volume), 2 = Moderate (affecting 26% to 50% of the lung volume), 3 = Severe (affecting 51% to 100% of the lung volume) where higher scores indicated more severity. The score of each participant was averaged over all 4 levels and both sides of lung. Mean score across 4 levels and both lungs = (Mean score across X levels for left lung + Mean score across X levels for right lung)/2. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study), Month 102 for adults and Month 84 for pediatrics
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 4 | 5
score on a scale
  Ground Glass Appearance | -1.21 (0.94) | -0.42 (0.41)
  Interstitial Lung Disease | -1.66 (1.20) | -1.35 (1.27)
  Pleural Thickening | 0 (0) | 0 (0)
  Reticulo-nodular Density | -2.19 (1.07) | -1.20 (1.30)

19. Secondary Outcome: Percent Change From Baseline in Percent Predicted Diffusing Capacity of Lungs For Carbon Monoxide (DLco) (Hemoglobin-Adjusted) at Month 78 for Adults and Month 84 for Pediatrics
Description: DLco was used to measure gas exchange across the alveolocapillary membrane. Percent predicted hemoglobin-adjusted DLco was calculated as: 100 x Adjusted DLco/Predicted DLco in unit of mL co/minute (min)/mmHg where, adjusted DLco = Observed DLco (in mL co/min/mmHg) divided by Hemoglobin-adjusted factor. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study), Month 78 for adults and Month 84 for pediatrics
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5 | 5
percent change | 55.29 (48.08) | 46.20 (48.46)

20. Secondary Outcome: Percent Change From Baseline in Platelet Count at Month 90 for Adults and Month 78 for Pediatrics
Description: Blood samples were collected at specified timepoints for the estimation of platelet count as ASMD is known to result in hematologic disorders. Baseline was defined as the average of all available values before the start of first infusion from original study
Time Frame: Baseline (Day 1 of original study), Month 90 for adults (pre-infusion) and Month 78 for pediatrics (pre-infusion)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 4 | 5
percent change | 21.83 (17.89) | 63.97 (32.67)

21. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein at Month 90 for Adults and Month 66 for Pediatrics
Description: Blood samples were collected at specified timepoints for fasting lipids as ASMD leads to progressive accumulation of lipids. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study), Month 90 for adults and Month 66 for pediatrics
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 4 | 5
percent change | -24.51 (11.05) | -37.30 (15.68)

22. Secondary Outcome: Participants From Adult Study DFI13412: Change From Baseline in Brief Fatigue Inventory (BFI) Questionnaire at Month 78
Description: The BFI involves a total of 9 items:3 of which measure BFI-fatigue severity score and 6 of which measure BFI-fatigue interference score. Score for each item measuring severity score is assessed by numerical rating scale (NRS); ranges from 0-10 from 0 (no fatigue) to 10 (worst imaginable fatigue) ultimately leading to overall severity score that ranges from 0-30. Respectively, amount that fatigue interfered with different aspects of participant's life during preceding 24 hours (general activity,mood,walking ability,normal work,relations with other people,and enjoyment of life) is captured as part of interference score.These different aspects are measured in scores ranging from 0:does not interfere and 10:completely interferes,ultimately leading to overall interference score ranging between 0-60. Higher scores in both categories mentioned below indicate worse outcome; mean is presented. Baseline was defined as last available non-missing value prior to first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 78
Population: Results are based on the Safety analysis set which consisted of all enrolled participants who received at least 1 infusion (partial or total) of olipudase alfa in the current study. Only those participants with data collected at specified timepoints for each specified category are reported.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults)
Number analyzed (Participants) | 5
score on a scale
  BFI-Fatigue Severity Scale Score | -0.9 (1.92)
  BFI-Fatigue Interference Scale Score | 0.6 (2.91)

23. Secondary Outcome: Participants From Adult Study DFI13412: Change From Baseline in Brief Pain Inventory-Short Form (BPI-SF) Questionnaire at Month 78
Description: The BPI-SF is a 15-item, validated, self-administered questionnaire designed to measure participant's perceived level of pain. The BPI-SF measured the participant's intensity of pain (sensory dimension), the interference of pain in participant's life (reactive dimension), and asked participant about pain relief, pain quality, and perception of cause of pain. Scoring was based on 4 out of 8 questions in pain severity domain, and 7 questions in pain interference domain, which used numerical rating scale. Pain severity response ranged from 0 = "No pain" to 10 = "Pain as bad as you can imagine". Pain interference response ranged from 0 = "Does not interfere" to 10 = "Completely interferes". Scores were averaged and mean is presented here. Higher scores indicated greater intensity of pain. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 78
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults)
Number analyzed (Participants) | 5
score on a scale
  BPI-SF: Pain Severity Scale Score | -1.5 (1.74)
  BPI-SF: Pain Interference Scale Score | 0.7 (3.13)

24. Secondary Outcome: Participants From Adult Study DFI13412: Change From Baseline in Chronic Respiratory Disease Questionnaire Self-Administered Standardized (CRQ-SAS) at Month 78
Description: The CRQ-SAS is a validated, self-administered questionnaire designed to evaluate health related quality of life (HRQoL) in adults with chronic airflow limitation, chronic respiratory disease and cystic fibrosis. It had 20 items and evaluated 4 dimensions of respiratory impairment (dyspnea, emotional function, fatigue and participant's feeling of control over the disease [mastery]). Each domain was measured on 7-point-scale, with 8 reserved for "not done" (1: worst and 7: best). Each domain score was calculated separately. Scores for each question of each domain were added together and divided by number of questions answered in each domain. Only items answered were scored. Mean of average score of completed items is reported. Higher scores indicated better HRQoL in each domain. Baseline was defined as last available non-missing value prior to first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 78
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Olipudase Alfa: Participants continued to receive olipudase alfa at the same dose as at the completion of original study-DFI13412 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible.
Arm/Group | Olipudase Alfa
Number analyzed (Participants) | 5
score on a scale
  Dyspnea Scale Score | 0.3 (0.59)
  Emotional Function Scale Score | 0.2 (1.49)
  Fatigue Scale Score | 0.3 (0.82)
  Mastery Scale Score | -0.5 (0.91)

25. Secondary Outcome: Participants From Pediatric Study DFI13803: Change From Baseline in Pediatric Quality of Life (PedsQL) Generic Core Total Scale Score at Month 72
Description: PedsQL included a child self-report for participants 5 to 18 years and parents' report of participants from 2 to 18 years. Child-reported: 23-item PedsQL Generic Core Scales report included 4 scales, physical functioning, emotional functioning, social functioning, and school functioning. Parent-reported: 21-item PedsQL Generic Core Scales report and included similar scales as above. Each item used a 5-point rating scale (from 0=never to 4=almost always). Items are reverse scored and linearly transformed to a 0 (almost always) -100 (never) scale. All summary/total scores were mean of specific items where higher score indicated better HRQoL. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5
score on a scale
  Child-reported | 10.4 (19.4)
  Parent-reported | 14.6 (20.1)

26. Secondary Outcome: Participants From Pediatric Study DFI13803: Change From Baseline in Difference Between Bone Age and Actual Age of Participants at Month 72
Description: Hand X-ray was performed on participant's left hand, fingers and wrist to assess the bone age. The X-rays were collected and read centrally by a third party blinded to participant number and study visit. At each visit, difference between the bone age and actual age at that visit was calculated. Difference in age in months was calculated as bone age in months minus real age at time of assessment in months. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: month
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5
month | 28.34 (24.68)

27. Secondary Outcome: Participants From Pediatric Study DFI13803: Change From Baseline in Height Z-score at Month 72
Description: Linear growth in pediatric participants was assessed by height Z-scores. Height Z-score, i.e., the height-for-age Z-score, is the number of standard deviations of the actual height of a child from the median height of the children of the corresponding age and sex as determined from the standard sample. A height Z-score of 0 is equal to the median and is considered normal. Negative numbers indicate values lower than the median and positive numbers indicate values higher than the median. For analysis, mean Z-score was calculated and an increase of mean height Z-score from baseline indicated an improvement on growth. Baseline was defined as the last available non-missing value prior to the first infusion in original study.
Time Frame: Baseline (Day 1 of original study) and Month 72
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
Number analyzed (Participants) | 5
Z-score | 2.31 (1.34)

ADVERSE EVENTS:
Time Frame: From the signature of informed consent up to 9 years or until olipudase alfa was commercially accessible, whichever came first
Description: Results are based on the Safety analysis set.
Groups:
- Olipudase Alfa: Participants From DFI13412 (Adults): Participants continued to receive olipudase alfa at the same dose as at the completion of original study-DFI13412 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible.
- Olipudase Alfa: Participants From DFI13803 (Pediatrics): Participants continued to receive olipudase alfa at the same dose as at the completion of original study-DFI13803 (up to 3.0 mg/kg) via IV infusion every 2 weeks for 9 years, or until olipudase alfa was commercially accessible, whichever came first, unless the participant decided to enter another olipudase alfa clinical trial within the 9-year period prior to when olipudase alfa was commercially accessible. During the study, pediatric participants who reached adult age (18 years old) received the adult infusion volume.
Arm/Group | Olipudase Alfa: Participants From DFI13412 (Adults) | Olipudase Alfa: Participants From DFI13803 (Pediatrics)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/5 | 10/20
Other Adverse Events (participants affected / at risk) | 5/5 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olipudase Alfa: Participants From DFI13412 (Adults) (N=5) | Olipudase Alfa: Participants From DFI13803 (Pediatrics) (N=20)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Otitis Media (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Craniofacial Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull Fractured Base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (3)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1)
Nuchal Rigidity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Poor Venous Access (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olipudase Alfa: Participants From DFI13412 (Adults) (N=5) | Olipudase Alfa: Participants From DFI13803 (Pediatrics) (N=20)
Pyrexia (General disorders) | 4 (97) | 18 (98)
Contusion (Injury, poisoning and procedural complications) | 4 (55) | 9 (148)
Headache (Nervous system disorders) | 5 (178) | 13 (91)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2022-04-15): https://cdn.clinicaltrials.gov/large-docs/04/NCT02004704/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT02004704/SAP_001.pdf